CLINICAL TRIAL: NCT05491239
Title: Optimal Postoperative Pain Management After Lung Surgery (OPtriAL): Multi-centre Randomised Trial
Brief Title: Optimal Postoperative Pain Management After Lung Surgery (OPtriAL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maxima Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Amsterdam UMC (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Louisa Spaans, Coordinating Investigator, MD, Maxima Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL75375.041.20
Record Dates: First submitted 2022-08-02; First posted 2022-08-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer; Pain, Postoperative; VATS; Locoregional Anaesthesia; Thoracic Epidural
MeSH Terms: conditions — Lung Neoplasms; Pain, Postoperative | interventions — Tea

STUDY DESIGN:
Intervention Model Description: This is a multi-centre randomised three-arm trial comparing continuous PVB, single-shot ICNB and TEA in a 1:1:1 ratio in patients who will undergo a VATS anatomic lung resection. We use a non-inferiority design with respect to the outcome measure 'pain' and a concomitant superiority design regarding 'quality of recovery'.
Masking Description: As the analgesic strategies highly differ in nature (with or without percutaneous catheter) and/or postoperative care (mobility with or without prerequisites, urinary catheter placement), blinding for the randomised strategy is unfeasible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thoracic epidural analgesia (Active Comparator): See intervention description
  Interventions: Procedure: Thoracic epidural analgesia
- Continuous regional paravertebral block (Experimental): See intervention description
  Interventions: Procedure: Continuous regional paravertebral block
- Single shot intercostal nerve block (Experimental): See intervention description
  Interventions: Procedure: Single shot intercostal nerve block

INTERVENTIONS:
Procedure: Thoracic epidural analgesia — After correct placement of the epidural catheter, a local anaesthetic (ropivacaine, levobupivacaine or bupivacaine) will be started and, according to in house protocols, an opioid will be added to the epidural solution. A provisional stop of the administration of the epidural infusion is planned after 48 hours (on the second postoperative day).
  Arms: Thoracic epidural analgesia
Procedure: Continuous regional paravertebral block — The PVB catheter is placed under general anaesthesia at the beginning of the VATS procedure under direct thoracoscopic vision. The level of the PVB catheter placement is chosen at the intercostal space of the largest incision (mostly thoracic level 4 or 5). Under direct thoracoscopic vision, the surgeon inserts a Touhy needle. The tip of the needle is observed beneath the pleural surface thoracoscopically. Injection of about 2 mL ropivacaine 7.5mg/mL will create subpleural hydrodissection to reach the adequate paravertebral plane for placement of the catheter. The PVB catheter is subsequently placed under direct thoracoscopic vision and left next to the sympathetic chain in the paravertebral space. Next, a bolus of ropivacaine (total amount 20 mL including the given amount for hydrodissection) is given through the catheter.
  Postoperatively, a ropivacaine 2 mg/mL pump for continuous infusion is given with an infusion rate of 8-14 ml/hour.
  Arms: Continuous regional paravertebral block
Procedure: Single shot intercostal nerve block — At the end of the surgery a single shot ICNB will be placed at 9 levels (thoracic level 2 to 10) with 2-3mL local anaesthetics per intercostal space under direct thoracoscopic vision. The injection site will be chosen just lateral from the sympathetic trunk. This group will have no analgesic catheters for continuous analgesia. No mobility restrictions are instructed in this group.
  Arms: Single shot intercostal nerve block

SUMMARY:
Adequate pain control after video-assisted thoracoscopic surgery (VATS) for lung resection is important to improve postoperative mobilisation, recovery, and to prevent pulmonary complications. So far, no consensus exists on optimal postoperative pain management after VATS anatomic lung resection.

Thoracic epidural analgesia (TEA) is the reference standard for postoperative pain management following VATS. Although the analgesic effect of TEA is clear, it is associated with patient immobilisation, bladder dysfunction and hypotension which may result in delayed recovery and longer hospitalisation. These disadvantages of TEA initiated the development of unilateral regional techniques for pain management. The most frequently used techniques are continuous paravertebral block (PVB) and single-shot intercostal nerve block (ICNB).

The investigators hypothesize that using either PVB or ICNB is non-inferior to TEA regarding postoperative pain and superior regarding quality of recovery (QoR). Signifying faster postoperative mobilisation, reduced morbidity and shorter hospitalisation, these techniques may therefore reduce health care costs and improve patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* Patients referred for anatomic lung resection (pneumonectomy, (bi)lobectomy or segmentectomy for either benign or malignant disease) with the intention of performing it by video-assisted thoracoscopic surgery (VATS) or robot-assisted thoracoscopic surgery (RATS)
* Patients should be able to provide informed consent and fill out questionnaires in Dutch language.

Exclusion Criteria:

* Patients with contra-indications for TEA or PVB (infection at skin site, increased intracranial pressure, non-correctable coagulopathy, bridging indication for therapeutic anticoagulation (CHADS-VASc ≥ 8), sepsis and mechanical spine obstruction) or allergic reactions to local anaesthetics will be excluded.
* Patients chronically using opioids for reasons not related to the operation will be excluded from the study since postoperative baseline opioid requirement will be higher and TEA remains the preferred technique for these patients.
* In case the lung surgeon estimates the operation to be performed through a thoracotomy instead of VATS/RATS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Pain scores | Postoperative day 0-2
  Proportion of pain scores ≥4 as assessed by the numerical rating scale (NRS) (measured from 0 until 10; lowest value signifying no pain and highest value signifying worst pain)
Quality of Recovery (QoR) | Postoperative day 1-2
  QoR measured with the QoR-15 questionnaire on postoperative 1 and 2 (maximum score of 150, the higher the score the better the outcome)

SECONDARY OUTCOMES:
cumulative use of opioids and analgesics | Postoperative day 0 until 3 as well as the use and dosage of opioid use at the follow-up period 2-3 weeks after the operation
  total opioid and non-opioid consumption as supplementary analgesic requirement
postoperative complications | until 2-3 weeks of follow-up
  according to the Clavien-Dindo classification;
hospitalisation | 30 postoperative days
  defined as the total number of days in hospital after the surgical intervention (including readmissions within the first 30 postoperative days), the following standardised discharge criteria after surgery will be applied in all participating hospitals: normal intake of nutrition, independent mobility, absence of fever (<38 °C), and no presence of chest tube;
patient satisfaction | Postoperative day 0 until 3
  5-point Likert scale: not at all satisfied, slightly satisfied, neutral, very satisfied and extremely satisfied
degree of mobility | Postoperative day 0 until 3
  4-point scale: on the bed (1), to the chair (2), to the toilet (3), outside the patient's hospital room(4)

CONTACTS AND LOCATIONS:
Locations (1):
- Maxima MC, Veldhoven, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will become available for non-commercial scientific research (open access) after a period of 12 months after the last data collection. Data request can be done by contacting the PI.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Spaans LN, Dijkgraaf MGW, Susa D, de Loos ER, Mourisse JMJ, Bouwman RA, Verhagen AFTM, van den Broek FJC; OPtriAL Study Group; Meijer P, Kuut M, Hanneman N, Bousema J, Franssen A, Brokx H, van Duyn E, Potters JW, van den Broek R, van Brakel T, Rijna H, Boom A, Noyez V, Hendriks JMH, Yogeswaran SK, Dickhoff C, van Dorp M. Intercostal or Paravertebral Block vs Thoracic Epidural in Lung Surgery: A Randomized Noninferiority Trial. JAMA Surg. 2025 Aug 1;160(8):855-864. doi: 10.1001/jamasurg.2025.1899. PMID 40560556
- [Derived] Spaans LN, Dijkgraaf MGW, Meijer P, Mourisse J, Bouwman RA, Verhagen AFTM, van den Broek FJC; OPtriAL study group. Optimal postoperative pain management after VATS lung resection by thoracic epidural analgesia, continuous paravertebral block or single-shot intercostal nerve block (OPtriAL): study protocol of a three-arm multicentre randomised controlled trial. BMC Surg. 2022 Sep 4;22(1):330. doi: 10.1186/s12893-022-01765-y. PMID 36058900

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-10-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT05491239/SAP_000.pdf